CLINICAL TRIAL: NCT05472428
Title: Autologous Bone Marrow Mononuclear Cell Administration in the Treatment of Neurologic Sequela in Children With Spina Bifida
Brief Title: Outcomes of Autologous Bone Marrow Mononuclear Cell Administration in the Treatment of Neurologic Sequelea in Children With Spina Bifida
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vinmec Research Institute of Stem Cell and Gene Technology (Other)
Collaborators: Vinmec Health Care System (Vingroup Joint Stock Company) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS. ĐT.19H1
Record Dates: First submitted 2022-07-09; First posted 2022-07-25 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Stem Cell Infusion
Keywords: Spina bifida; mononuclear cell; neurologic sequelea
MeSH Terms: conditions — Spinal Dysraphism

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Autologous BMMNC transplantation (Experimental): - Autologous bone marrow mononuclear cell transplantation 2 intrathecal administrations of autologous bone marrow mononuclear cells at baseline and 6 months afterward
  Interventions: Combination Product: Autologous bone marrow mononuclear cell transplantation

INTERVENTIONS:
Combination Product: Autologous bone marrow mononuclear cell transplantation — Transplantation of Autologous Bone Marrow Mononuclear cells

SUMMARY:
The aim of this study was to evaluate the safety and efficacy of autologous bone marrow mononuclear cell infusion in the management of neurological sequelae in children with spina bifida

DETAILED DESCRIPTION:
The aim of this study was to evaluate the safety and effectiveness of autologous bone marrow mononuclear cells in 11 patients with spina bifida at Vinmec Research Institute of Stem Cell and Gene Technology in Hanoi, Vietnam from 2016 to 2020

ELIGIBILITY:
Inclusion Criteria:

* The patient who was diagnosed with lumbar spina bifida underwent spinal cord close-up surgery.
* Both genders.
* Aged between 6 months and 15 years old.
* Exhibited bowel disorders (constipation, fecal incontinence) and urinary dysfunction (urinary retention or leakage).

Exclusion Criteria:

* Vertebrae clefts in the chest, neck, and other spinal locations.
* Coagulopathy.
* Acute and chronic infection.
* Kidney function disorder, liver failure
* Patients with complex cardiovascular diseases (including valvular heart disease, cardiomyopathy, arrhythmia, congenital heart disease, hypertrophy syndrome).
* Distress

Ages: 6 Months to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 11 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2020-12-25 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Adverse events and serious adverse events | up to the 12-month period following treatment
  Incidence of the adverse events or serious adverse events after infusion

SECONDARY OUTCOMES:
Bristol stool scale | up to the 12-month period following treatment
  The Bristol stool scale comes in 7 types: Type 1-2 indicate constipation; type 3-4 are ideal stools as they are easier to pass; type 5-7 may show diarrhea and urgency.
Rectoanal inhibitory reflex | up to the 12-month period following treatment
  The rectoanal inhibitory reflex (RAIR) is a reflex characterized by transient involuntary relaxation of the internal anal sphincter in response to distention of the rectum with the normal value <= 14.7 ml
Bladder sensation | up to the 12-month period following treatment
  The cystometry was used to assess bladder sensation
Urinary retention | up to the 12-month period following treatment
  urinary retention is assessed via cytometry
Urinary incontinence | up to the 12-month period following treatment
  Urinary incontinence is assessed via cytometry
Lower limb motor functions | up to the 12-month period following treatment
  Lower limb motor function was assessed via manual muscle testing (MMT)

CONTACTS AND LOCATIONS:
Overall Officials: Liem T Nguyen, MD., PhD, Principal Investigator — Vinmec Research Institute of Stem Cell and Gene Technology
Locations (1):
- Vinmec Research Institute of Stem Cell and Gene Technology, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Liem NT, Chinh VD, Thinh NT, Minh ND, Duc HM. Improved Bowel Function in Patients with Spina Bifida After Bone Marrow-Derived Mononuclear Cell Transplantation: A Report of 2 Cases. Am J Case Rep. 2018 Aug 25;19:1010-1018. doi: 10.12659/AJCR.909801. PMID 30143601
- [Result] Aghayan HR, Arjmand B, Yaghoubi M, Moradi-Lakeh M, Kashani H, Shokraneh F. Clinical outcome of autologous mononuclear cells transplantation for spinal cord injury: a systematic review and meta-analysis. Med J Islam Repub Iran. 2014 Oct 14;28:112. eCollection 2014. PMID 25678991
- [Derived] Than UTT, Nguyen LT, Nguyen PH, Nguyen XH, Trinh DP, Hoang DH, Nguyen PAT, Dang VD. Inflammatory mediators drive neuroinflammation in autism spectrum disorder and cerebral palsy. Sci Rep. 2023 Dec 18;13(1):22587. doi: 10.1038/s41598-023-49902-8. PMID 38114596
- [Derived] Nguyen LT, Le HT, Nguyen KT, Bui HT, Nguyen APT, Ngo DV, Hoang DM, Ngo MD. Outcomes of autologous bone marrow mononuclear cell administration in the treatment of neurologic sequelae in children with spina bifida. Stem Cell Res Ther. 2023 Apr 28;14(1):115. doi: 10.1186/s13287-023-03349-w. PMID 37118832